CLINICAL TRIAL: NCT05487950
Title: Rivaroxaban Versus Standard of Care for Patients With Excessive Atrial Ectopy or Short Atrial Runs and High Embolism Risk
Acronym: SHORT RUN AF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200002
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Excessive Supraventricular Ectopies or Short Atrial Runs (ESVEA)
Keywords: atrial fibrillation; RIVAROXABAN; embolism; short atrial runs (ESVEA)
MeSH Terms: conditions — Atrial Fibrillation; Embolism

STUDY DESIGN:
Intervention Model Description: This is a phase III prospective superiority randomized open-label multicenter study with 2 parallel groups (control vs. experimental group).
  Our study will test the superiority of anticoagulation treatment with Rixaroxaban (experimental group) compared to SOC (control group).
  This is a phase III prospective superiority randomized, open-label multicenter study with 2 parallel groups (control vs. experimental group).
  Patients with excessive supraventricular ectopies or short atrial runs (ESVEA) defined as ≥ 1% PAC /24 hours or any atrial runs ≥ 20 PACs on a 24-hour Holter ECG monitoring and CHA2DS2VASC score ≥ 3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Patients in the Rivaroxaban group will receive Rivaroxaban at the dose of 15 mg once daily ((or 10 mg if renal insufficiency) during 2 years.
  Interventions: Drug: Rivaroxaban group
- group control (No Intervention): Patients in the control group will be followed according to the standard of care (SOC) chosen by the investigator during 2 years. Additions or changes to SOC are allowed during the patient participation in the study based on patient status and evolution (with the exception of the use of anticoagulant therapy).

INTERVENTIONS:
Drug: Rivaroxaban group — Patients assigned in the Rivaroxaban group will receive 15 mg once day or 10 mg if dosage modification is needed due to renal insufficiency (Creatinine clairance calculated with the Cockroft formula between 30 or 49 ml/min).
  Arms: experimental group

SUMMARY:
The primary objective of the Short Run AF study is to evaluate the efficacy and safety of long term anticoagulation with rivaroxaban against standard of care (SOC) in patients with ESVEA and CHA2DS2VASC score ≥3 on the incidence of ischemic stroke and peripheral embolism after 2 years follow-up and the occurrence of major bleeding events.

The primary efficacy endpoint is the first ischemic stroke or peripheral embolism detected clinically and on systematic cerebral MRIs in a time-to-event analysis.

The primary safety outcome is major bleeding at any site in the body according to the criteria of the International Society of Thrombosis and Hemostasis (ISTH)(23-25).

DETAILED DESCRIPTION:
Patients with atrial fibrillation (AF) (> 30 consecutive seconds of arrhythmia) and high risk embolism meaning CHA2DS2VASC score ≥2 are candidate for long term oral anticoagulation. In addition, patients with excessive supraventricular ectopies or short atrial runs (ESVEA) but no documented AF are also at higher risk of systemic embolism compared to normal population. ESVEA is a frequent clinical situation observed approximately in up to 15% on systematic 24-hour Holter ECG in patients over 65 years old with cardiovascular risk factors. In addition, it is associated with a higher risk of peripheral arterial thromboembolism. However, it remains unclear if this former population could benefit from long-term oral anticoagulation.

To date no other studies have evaluated the effect of anticoagulation for patients with excessive atrial ectopies or short atrial runs. Also, to our knowledge, no study evaluating this problematic is ongoing. This population is actually not treated but in real clinical practice, patients with high CHA2DS2VASC score presenting with ESVEA could be candidate for oral anticoagulation. If it is demonstrated that patients with ESVEA and CHA2DS2VASC score ≥ 3 could benefit from oral anticoagulation and particularly new oral anticoagulants, it would change the everyday practice of cardiologist or gerontologist.

Our hypothesis is that long term anticoagulation with rivaroxaban could reduce drastically (50%, comparable with its effect during AF) the incidence of stroke or other thromboembolism events compared to standard of care (SOC), with a possible but moderate increased risk of bleeding compared to SOC that should remain acceptable compared to the reduction of stroke (net clinical benefit).

In this study, the study also attempt to describe the clinical course of patients with ESVEA in terms of global cardiovascular events, occurrence of documented atrial fibrillation or cognitive decline with an everyday practice follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years old
* Diagnosis of excessive supraventricular ectopy activity defined as ≥ 1% PAC / 24 h or any atrial runs ≥ 20 PACs on a 24-hour Holter ECG monitoring (the indication for the Holter will be let at the discretion of the doctor according to international guidelines indication)
* High risk embolism defined by a CHA2DS2VASC score ≥ 3
* Written consent from patient
* Patients able to attend consultations and Cerebral MRI at baseline and 24 months at the participating centre.
* Ability to understand and comply with the study protocol
* Affiliation of social security regime

Exclusion Criteria:

* According to the SmPC, any contraindication to Rivaroxaban (particularly patients with ongoing major bleeding, vascular complication, prior haemorrhagic stroke or over recent stroke) or one of its excipients.
* Inability to perform cerebral MRI
* Life expectancy <24 months
* History of major hemorrhage after taking Rivaroxaban
* Documented atrial fibrillation or any other indication for oral anticoagulation
* Patients with previous documented AF
* Valvular congenital heart disease
* Anticoagulant agents in the month prior to the inclusion visit
* Acute coronary syndrome, coronary revascularization (percutaneous coronary intervention or coronary artery bypass surgery) or in the past 30 days
* Requires long-term antiplatelet therapy other than aspirin (i.e., patient requires any platelet aggregation inhibitor in addition to study treatment, in particular, the combination of two platelet aggregation inhibitors)
* Ongoing need for strong inhibitors of both CYP3A4 and P-glycoprotein (e.g., ketoconazole, itraconazole, ritonavir or clarithromycin)
* Ongoing need for strong inducers of both CYP3A4 and P-glycoprotein (e.g., rifampin, carbamazepine, phenytoin)
* Participants considered by the investigator to be unsuitable for the study for any of the following reasons:Patient refuse the treatment with rivaroxaban or anticipated to have poor compliance on study drug treatment or Unwilling to attend study follow-up visits
* Cancer or other life threatening conditions
* Severe, disabling stroke within the previous 6 months, or any stroke within the previous 14 days
* Conditions associated with an increased risk of bleeding:

  1. Major surgery within the previous month
  2. Planned surgery or intervention within the next 3 months
  3. History of intracranial, intraocular, spinal, retroperitoneal or atraumatic intra-articular bleeding
  4. Gastrointestinal hemorrhage within the past year
  5. Symptomatic or endoscopically documented gastroduodenal ulcer disease in the previous 30 days
  6. Hemorrhagic disorder or bleeding diathesis
  7. Need for anticoagulant treatment of disorders other than atrial fibrillation
  8. Fibrinolytic agents within 48 hours of study entry
  9. Uncontrolled hypertension (systolic blood pressure greater than 180 mm Hg and/or diastolic blood pressure greater than 100 mm Hg)
  10. Recent malignancy or radiation therapy (within 6 months) and not expected to survive 3 years
* Severe renal impairment (estimated creatinine clearance <30 mL/min or less)
* Active infective endocarditis
* Active liver disease, including but not limited to, associated or not with coagulopathy and a clinically significant risk of bleeding, including cirrhotic patients with a Child Pugh class B or C score.
* Persistent ALT, AST, Alk Phos greater than twice the upper limit of the normal range
* Known active hepatitis C (positive HCV RNA)
* Known active hepatitis B (HBs antigen +, anti HBc IgM +)
* Known active hepatitis A
* Anemia (hemoglobin level less than 110 g/L) or thrombocytopenia (platelet count less than 150 X 109/L)
* Patients who have received an investigational drug in the past 30 days
* Patients considered unreliable by the investigator, or having any condition which, in the opinion of the investigator, would not allow safe participation in the study (e.g., drug addiction, alcohol abuse)
* Patient with cardiac prosthetic devices : Reveal, pace-maker, automatic implantable defibrillator
* Participation in another interventional clinical trial
* Patient on AME (state medical aid)
* Persons under psychiatric care
* Adults subject to a legal protection measure (guardianship, curatorship and safeguard of justice)Patients deprived of their liberty by a judicial or administrative decision

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-04-05 (Estimated); Primary Completion 2027-04-05 (Estimated); Study Completion 2027-04-05 (Estimated)

PRIMARY OUTCOMES:
incidence of first ischemic stroke or peripheral embolism | during 28 months follow-up
  The primary efficacy endpoint is the first ischemic stroke or peripheral embolism detected clinically and on systematic cerebral MRIs in a time-to-event analysis.
incidence of major bleeding at any site in the body | 2-year follow-up.
  The primary safety outcome is major bleeding at any site in the body according to the criteria of the International Society of Thrombosis and Hemostasis (ISTH)(23-25).

SECONDARY OUTCOMES:
the incidence of documented atrial fibrillation | 2-year follow-up.
  the incidence of documented atrial fibrillation diagnosed from patient symptoms or systematic 24 hours ECG Holter performed at 2-year follow-up.

IPD SHARING:
Plan to Share IPD: No